CLINICAL TRIAL: NCT02525432
Title: A Multicenter Trial of Autologous Bone Marrow Mononuclear Cells for the Treatment of Adult Severe Traumatic Brain Injury
Brief Title: Autologous Stem Cell Study for Adult TBI (Phase 2b)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Principal Investigator, Charles Cox, Professor, Department of Pediatric Surgery, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC-MS-16-0283
Record Dates: First submitted 2015-03-23; First posted 2015-08-17 (Estimated); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Brain Injuries, Traumatic; Brain Injuries, Acute; TBI (Traumatic Brain Injury)
Keywords: Mesenchymal Stromal Cells, Multipotent; Multipotent Mesenchymal Stromal Cells; Stem Cells, Mesenchymal
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Autologous BMMNC Infusion (Experimental): Subjects randomized to the treatment group will undergo a bone marrow harvest and then receive an autologous infusion of BMMNC's starting with the lowest dose (6 x 10^6 cells/kg body weight) and progressing to the high dose of 9 x 10^6 cells/kg body weight using a Bayesian adaptive dose escalation design.
  Interventions: Biological: Autologous BMMNC Infusion
- Placebo Infusion (Placebo Comparator): Subjects randomized to the placebo control group will undergo a "sham" bone marrow harvest.
  Interventions: Biological: Placebo Infusion

INTERVENTIONS:
Biological: Placebo Infusion — In addition to the standard of care provided to all patients with traumatic brain injury, subjects assigned to the placebo control group will undergo a sham bone marrow harvest and receive a placebo infusion of saline.
  Arms: Placebo Infusion
Biological: Autologous BMMNC Infusion — In addition to the standard of care provided to all patients with traumatic brain injury, subjects assigned to the BMMNC treatment group will undergo a bone marrow harvest and then receive an autologous stem cell infusion.
  Other Names: Stem Cell Infusion
  Arms: Autologous BMMNC Infusion

SUMMARY:
The purpose of this study is to determine the effect of intravenous infusion of autologous bone marrow mononuclear cells (BMMNC) on brain structure and neurocognitive/functional outcomes after severe traumatic brain (TBI) injury in adults. The primary objective is to determine if the intravenous infusion of autologous BMMNC after severe TBI results in structural preservation of global gray matter (GM) volume and white matter (WM) volume and integrity; as well as select regions of interest in the corpus callosum. THe secondary objectives are to determine if autologous BMMNC infusion improves functional and neurocognitive deficits in adults after TBI; reduces the neuroinflammatory response to TBI; evaluate spleen size and splenic blood flow over time using ultrasound and corresponding changes in inflammatory cytokines; and infusion related toxicity and long-term follow-up safety evaluations.

DETAILED DESCRIPTION:
Traumatic brain injuries are associated with 33% of all trauma related deaths. There are no effective therapies to treat secondary brain injury and the post-injury response of CNS apoptosis and neuroinflammation. Pre-clinical and Phase I clinical progenitor cell therapies have shown promise in TBI/stroke via (1) promotion of CNS structural preservation, and (2) reducing the neuroinflammatory response to injury.

This is a multicenter, randomized, blinded, Bayesian CRM dose-escalation placebo-controlled study designed to treat severe, acute TBI in adult patients with an IV infusion of autologous bone marrow mononuclear cells. 55 adult TBI patients will be randomized to receive a single IV infusion of BMMNs (6 x 10^6 or 9 x 10^6) or placebo.

Study subjects will be consecutive admissions of adults with severe TBI meeting inclusion/exclusion criteria. Adults, ages 18-55 years, hospitalized at Memorial Hermann Hospital (Houston, Texas) for severe TBI (GCS 3-8) will be screened for eligibility. Informed consent, the bone marrow/sham harvest, and stem cell/placebo infusion must take place within 48 hours of the initial injury.

Following consent and baseline procedures, subjects will be randomized in a 3:2 ratio (using permuted blocks and stratified by GCS of 3-4 or 5-8) to autologous BMMNC infusion (n=33) and placebo (n = 22), respectively. Administration will begin with the lowest dose (i.e. 6 x 10^6 cells/kg body weight) with each dose given to cohorts of 3 subjects treated with BMMNC (note: the cohort size refers only to subjects treated with autologous BMMNC). After each cohort of 3 subjects treated with autologous BMMNC infusion (accumulated on average after every 5.5 adults randomized), the dosage for the next cohort of 3 autologous BMMNC-treated subjects will be determined by the CRM based on the findings for all subjects previously treated and the prior probabilities of the likelihood of toxicity assigned by the investigators before starting the study. At all doses, the algorithm is designed to avoid administering doses that will have a p(toxicity) exceeding 0.15.

Subjects will be monitored closely for infusion related toxicity and complications during the first 14 days post-infusion while also receiving the usual standard of care for traumatic brain injury . Safety and outcome assessments will be performed at 1, 6, and 12 months post-injury study visits.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 to 55 years of age on the day of injury,
2. Non-penetrating closed head trauma.
3. Glasgow Coma Score between (GCS) between 3 and 8, (best un-medicated post-resuscitation score during screening).
4. Ability to obtain legally authorized representative consent for participation and complete the BMMNC/Sham harvest and cell/placebo infusion within 48 hours of the initial injury.
5. Ability to speak English or Spanish.

Exclusion Criteria:

1. Known history of:

   1. previous brain injury,
   2. intellectual deficiency or psychiatric condition likely to invalidate our ability to assess post-injury changes in cognition or behavior,
   3. neurologic impairment and/or deficit,
   4. seizure disorder requiring anti-convulsant therapy,
   5. recently treated significant infection,
   6. renal disease/altered renal function (post-resuscitation serum creatinine > 1.5 mg/dL),
   7. chronic hepatic disease or altered liver function (post-resuscitation SGPT > 150 U/L, and/or T. Bilirubin >1.3 mg/dL),
   8. cancer,
   9. Chemical or ETOH dependency,
   10. immunosuppression (admission WBC < 3X103),
   11. HIV positive status;
2. Obliteration of perimesencephalic cistern on initial head CT/MRI suggesting prolonged hypoxic ischemic insult;
3. Initial hospital ICP > 40 mm Hg;
4. Hemodynamic instability at the time of screening defined as SBP < 90mmHg, ongoing fluid resuscitation and/or requirement for inotropic support to maintain MAP at or above normals for age - does not include CPP based inotropic support;
5. Uncorrectable coagulopathy at the time of screening;
6. Unstable pelvic fractures that in the P.I.'s opinion would preclude the bone marrow / sham harvest;
7. Pulmonary contusions defined as a chest x-ray with non-anatomic opacification and PaO2:FiO2 ratio < 250 associated with the mechanism of injury;
8. Greater than AAST Grade III solid or hollow visceral injury of the abdomen and/or pelvis diagnosed by CT or other imaging;
9. Spinal cord injury diagnosed by CT or MR imaging or by clinical findings;
10. Persistent hypoxia defined as SaO2 < 94% for > 30 minutes occurring at any time from hospital admission to time of consent;
11. Positive pregnancy test (if applicable);
12. Concurrent participation in an interventional drug/device research study;
13. Unwillingness to return for follow-up visits;
14. Contraindications to MRI.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Macro and micro structural properties of grey matter (GM) and white matter (WM) regions will measured using high-resolution anatomical MRI and diffusion tensorm imaging and comparisons made between groups. | up to 6 months. Post Head Injury
  Subjects will undergo three 3T-MRI evaluations. The first will occur 7 to 10 days after hospitalization, when clinically stable. The following five pulse sequences constitute a complete imaging session: 1) conventional localizer/scout 2) 3D isotropic T1-weighted MPRAGE 3) 3D isotropic T2-weighted TSE 4) 32-direction single-shot spin-echo diffusion sensitized echo-planar (DTI-32dir) 5) 3D-FLAIR.
  The 3T-MRI will be repeated at 1 and 6 months post-injury. Composite scores will be calculated for comparison.

SECONDARY OUTCOMES:
Brain imaging measures of GM and WM structural integrity will be compared to functional and neurocognitive scores and comparisons made between groups. | Changes From Baseline to 6 mo. Post Head Injury
  Group differences in functional and neuropsychological outcomes will be assessed. Outcome scores will be correlated with specific macrostructural and microstructural metrics from the MRI. Composite scores will be calculated for comparison.
Compare neuro-inflammatory biomarkers between groups.. | Changes From Baseline to 6 mo. Post Head Injury
  CSF and plasma samples will be analyzed for neuro-inflammatory biomarkers and comparisons made between groups.
Measure the number of participants with infusion related adverse events. | up to 6 mo. Post Head Injury
  Infusion related adverse events will be determined from analysis of standard of care ICU monitoring data and comparisons made between groups.
Measure spleen ultrasound size over time and corresponding changes in inflammatory cytokines. | up to 6 mo. Post Head Injury
  Spleen ultrasound volume will be measured. A comparison of results between groups will help in understanding the contribution of the spleen in the systemic inflammatory responses after acute TBI.
Determine if microglial activation is associated with TBI and can be accurately measured with brain PET and DT-MRI imaging when compared to PET imaging data from healthy volunteers (enrolled under a different protocol). | 1 yr. Post Head Injury
  Brain PET and DT-MRI imaging will be obtained 1yr post injury. The outcome measures will be PET-MRI imaging SUV (standardized uptake values) based upon injected dose per patient weight. Voxel-wise analysis of regions of interest (ROI) will focus on: Midbrain, thalamus, hippocampus and cortical subdivisions which will be compared over time and to imaging data from healthy volunteers (enrolled under a different protocol). The SUV in ROIs will be correlated with a battery of functional outcomes measures focusing on the NINDS Common Data Elements. The degree of microglial activation will be correlated with the degree of volumetric loss in specific ROIs.
Quantify the extent and location of microglial activation by brain PET imaging and how activity correlates with performance of neurocognitive outcomes measures. | 1 yr. Post Head Injury
  Brain PET and DT-MRI imaging will be obtained 1yr post injury. The outcome measures will be PET-MRI imaging SUV (standardized uptake values) based upon injected dose per patient weight. Voxel-wise analysis of regions of interest (ROI) will focus on: Midbrain, thalamus, hippocampus and cortical subdivisions which will be compared over time and to imaging data from healthy volunteers (enrolled under a different protocol). The SUV in ROIs will be correlated with a battery of functional outcomes measures focusing on the NINDS Common Data Elements. The degree of microglial activation will be correlated with the degree of volumetric loss in specific ROIs.
Determine the extent to which an IV infusion of autologous BMMNC post-injury impacts microglial activation by brain PET imaging. | 1 yr. Post Head Injury
  Brain PET and DT-MRI imaging will be obtained 1yr post injury. The outcome measures will be PET-MRI imaging SUV (standardized uptake values) based upon injected dose per patient weight. Voxel-wise analysis of regions of interest (ROI) will focus on: Midbrain, thalamus, hippocampus and cortical subdivisions which will be compared over time and to imaging data from healthy volunteers (enrolled under a different protocol). The SUV in ROIs will be correlated with a battery of functional outcomes measures focusing on the NINDS Common Data Elements. The degree of microglial activation will be correlated with the degree of volumetric loss in specific ROIs.

CONTACTS AND LOCATIONS:
Overall Officials: Charles S Cox, MD, Principal Investigator — UTHealth McGovern Medical School, Houston, TX
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Data will be reported in aggregate.